CLINICAL TRIAL: NCT02220465
Title: Using Physical Activity to Reduce Smoking Cue Reactivity Among Low-Income Smokers Preparing to Quit Smoking
Brief Title: Step-up to Quit: Using Low-to-moderate Intensity Exercise for Reducing Smoking Cue Reactivity Among Low-income Smokers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13CRP14560028
Record Dates: First submitted 2014-08-15; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-01

CONDITIONS: Sedentary Lifestyle; Cigarette Smoking
Keywords: sedentary; smoking; cue reactivity; physical activity
MeSH Terms: conditions — Sedentary Behavior; Cigarette Smoking; Smoking; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA+ Smoking Cessation (LMPA) (Experimental): This intervention integrates low-to-moderate physical activity (PA) with evidence based smoking cessation programming. Over the 4-week treatment period, the intervention (1 in-person and 3 phone counseling sessions) focuses on (a) gradually increasing routine PA during the pre-quit period and maintaining PA post quit day (b) increasing daily PA (steps/day) using a weekly tailored algorithm with the goal of achieving 10,000 steps by Week 4 (quit day) and (c) training participants to use PA as a primary urge management strategy, thereby embedding PA within evidence-based smoking cessation counseling. Other components include additional smoking urge management skills, increasing motivation to quit, overcoming barriers and maintaining PA for quitting and staying smoke-free .
  Interventions: Behavioral: PA+ Smoking Cessation (LMPA)
- Standard Care Smoking Counseling (SCC) (Active Comparator): The control intervention parallels the format of the LMPA intervention with focus only on behavioral and cognitive urge management strategies (avoiding/escaping high-risk situations, stimulus control) and minimizing the probability that participants in the control group would increase increase/use PA during the intervention period. Participants are provided a pedometer without any instructions or encouragement around increasing walking/steps during the 8-week intervention period.
  Interventions: Behavioral: Standard Care Smoking Counseling (SCC)

INTERVENTIONS:
Behavioral: PA+ Smoking Cessation (LMPA)
  Arms: PA+ Smoking Cessation (LMPA)
Behavioral: Standard Care Smoking Counseling (SCC)
  Arms: Standard Care Smoking Counseling (SCC)

SUMMARY:
The study's primary aim is to test the hypothesis that an intervention that integrates low to moderate physical activity (walking) with evidence-based smoking cessation counseling (LMPA) will result is greater reductions in quit-day reactivity to smoking cues (a behavioral predictor of smoking relapse) as compared to standard care smoking cessation counseling (control group) in a sample of low-income sedentary male and female smokers. The study will also test the hypothesis that the participants randomized to the LMPA intervention will have greater quit rates at one-week and one-month post quit day follow ups.

DETAILED DESCRIPTION:
Tobacco use and lack of physical activity (PA) are preventable health behaviors contributing to disproportionate rates of morbidity/mortality (MM) among low income underserved adults. Comprehensive interventions incorporating treatment of multiple risk behaviors can have immense public health impact. The goal of this study is to improve uptake of PA during the pre-quit period by promoting low to moderate intensity PA (LMPA/walking) during the pre-quit preparatory period to promote smoking cessation among low-income sedentary smokers. Eligible participants (sedentary, >5 cigs/day) will be randomized to 8-week LMPA vs. standard of care (SCC) intervention. LMPA group intervention focuses on (a) increasing daily steps using a tailored algorithm with a goal of reaching 10,000 steps/day by Week 4 (quit day) and (b) integrates PA with evidence-based smoking cessation programming by explicitly linking short bouts of PA with urge management training during the pre-quit period. The SCC group receives standard care smoking cessation counseling. Group differences in quit day reduction (extinction) of smoking urge reactivity using an analog cue-exposure paradigm, and smoking quit rates at 1-week and 1-month follow-up will be examined.

ELIGIBILITY:
Inclusion Criteria:

* intent-to-treat sedentary male and female smokers (intention to quit within the next 6 months) - - - smoke 6 or more cigarettes per day.
* Sedentary critieria: not purposeful physical activity for less than 20 minutes of vigorous intensity, or less than 60 minutes of moderate intensity physical activity per week, or less than 100 minutes of time spent walking per week.

Exclusion Criteria:

* pregnancy
* current substance abuse (e.g., alcohol, cocaine, or stimulants);
* current diagnosis or treatment of bipolar and psychotic disorder (e.g., use of Haldol, Thorazine).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Smoking Cue Reactivity on Quit Day | 4-weeks
  smoking cue reactivity is a behavioral predictor of smoking outcomes. We anticipate that the LMPA intervention will experience greater reductions (extinction) during a controlled, massed cue exposure procedure on their quit day than the Standard care control (SCC) group.

SECONDARY OUTCOMES:
Quit rates at follow ups | 7 days prior to 1week and 1 month follow up assessments
  7-day point prevalence abstinence will be assessed using the 7-day timeline follow back administered at 1-week and 1-month follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Uma S Nair, PhD, Principal Investigator — Temple University
Locations (1):
- Temple university, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Nair US, Haynes P, Collins BN. Baseline sleep quality is a significant predictor of quit-day smoking self-efficacy among low-income treatment-seeking smokers. J Health Psychol. 2019 Sep;24(11):1484-1493. doi: 10.1177/1359105317740619. Epub 2017 Nov 15. PMID 29139311
- [Derived] Nair US, Patterson F, Rodriguez D, Collins BN. A telephone-based intervention to promote physical activity during smoking cessation: a randomized controlled proof-of-concept study. Transl Behav Med. 2017 Jun;7(2):138-147. doi: 10.1007/s13142-016-0449-x. PMID 27896797